CLINICAL TRIAL: NCT01164696
Title: A Prospective Observational Study to Evaluate Quality of Life and Costs in a Real Life Setting in Patients Treated With 90Y-Zevalin
Brief Title: A Prospective Observational Study to Evaluate the Quality of Life and the Costs in a Real Life Setting in Patients Who Are Treated With 90Y-Zevalin
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 13455; ZV0710BE
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Lymphoma, Follicular; Non-Hodgkin Lymphoma
Keywords: Quality of Life, Health Care Costs
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: [90]Y-ibritumomab tiuxetan (Zevalin, BAY86-5128)

INTERVENTIONS:
Drug: [90]Y-ibritumomab tiuxetan (Zevalin, BAY86-5128) — Zevalin was administered according to the directives in the approved package leaflet.

SUMMARY:
The objective of this study is to compare hematological toxicity, costs, health-related quality of Life (HR-QOL) and outcomes observed in real life in the Belgian Non-Hodgkin Lymphoma (NHL) population receiving 90Y-Zevalin, with model-predicted data at reimbursement on the basis of a clinical trial in heavily pre-treated NHL.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer of the lymph nodes of follicular type at study inclusion
* The patient has relapsed or has refractory disease, after previous treatment with rituximab
* Treating physician has decided to treat the patient with a 90Y-Zevalin regimen
* The patient is >= 18 years of age
* Patient has given informed consent

Exclusion Criteria:

* Patient is unwilling or unable to give informed consent
* Patient is participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with relapsed or refractory FL who have been treated with 90Y-Zevalin in Belgium within the first 24 months after ethics approval
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The medical resources consumed due to hematological adverse events that occurred following treatment with 90Y-Zevalin treatment | one year after inclusion

SECONDARY OUTCOMES:
the health related quality of life prior to and following treatment (using EQ-5D and FACT-LYM) | baseline: before 1st administration, 8 days after baseline, 1, 2 & 3 months after baseline
the clinical outcomes (survival status, response status), TTNT (time to next treatment) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Belgium